CLINICAL TRIAL: NCT00517556
Title: Continuous Administration of a Monophasic Oral Contraceptive in the Treatment of Primary Dysmenorrhea
Brief Title: Continuous Administration of Oral Contraceptive, Primary Dysmenorrhea
Acronym: Dysmenorrhea
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Richard S. Legro, M.D., Professor, Obstetrics and Gynecology and Public Health Sciences, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 25239
Record Dates: First submitted 2007-05-18; First posted 2007-08-17 (Estimated); Results first posted 2017-04-28 (Actual); Last update posted 2017-04-28 (Actual); Status verified 2017-03

CONDITIONS: Dysmenorrhea
Keywords: Dysmenorrhea; continuous OCP
MeSH Terms: conditions — Dysmenorrhea | interventions — Contraceptives, Oral

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- study group (CCOCP) (Experimental): treatment with monophasic oral contraceptive (gestodene 0,075 mg /ethinyl estradiol 20 mcg) for 168 continuous days through six cycles
  Interventions: Drug: CCOCP
- control group (traditional OCP) (Active Comparator): treatment with monophasic oral contraceptive (gestodene 0,075 mg /ethinyl estradiol 20 mcg) for traditional (21 active days/7 inactive days) regimen through six cycles.
  Interventions: Drug: Traditional OCP

INTERVENTIONS:
Drug: CCOCP — (CCOCP) continuous treatment with Monophasic oral gestodene/ethinyl estradiol
  Other Names: Oral contraceptives
  Arms: study group (CCOCP)
Drug: Traditional OCP — (traditional OCP) (21 active days/7 inactive days) treatment regimen
  Other Names: Oral contraceptives
  Arms: control group (traditional OCP)

SUMMARY:
The primary hypothesis is that continuous administration of an OCP (CCOCP regimen) will result in more pain relief than a traditional 21/7 administration in primary dysmenorrhea (PD) patients.

DETAILED DESCRIPTION:
It is well established that excess prostaglandin production in primary dysmenorrhea (PD) leads to ischemia of the uterine muscle, which consequently causes pelvic pain. A large number of drugs have been studied for pain relief in dysmenorrhea patients with non-steroid anti-inflammatory drugs (NSAIDs) being the most effective with the overall success rate of more than 75%. Oral contraceptive pills (OCP) are also an established treatment for PD with the success rate of 70%. Lately, OCP's have been used continuously in patients with endometriosis and had better pain control than traditional administration of OCP.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women ages 18-35 with a history of PD (onset < 3 years after menarche).
* Subjects must have had regular (25-31 day) menstrual cycles for the three month period preceding enrollment, with symptoms of moderate to severe PD during those cycles.

Exclusion Criteria:

* Patients who have contraindications to OCP therapy.
* Known or suspected secondary dysmenorrhea (major abdominal or pelvic surgery, endometriosis, pelvic inflammatory disease (PID), ovarian cysts, pathological vaginal secretion, chronic abdominal pain, inflammatory bowel disease, irritable bowel syndrome).
* Concomitant treatment with oral contraceptives, GnRH agonists and antagonists, antiandrogens, gonadotropins, anti-obesity drugs.
* The use of contraceptive implants, injectable contraceptives or intrauterine devices. The washout period on all these medications will be 3 months.
* Migraines, depression requiring hospitalization or associated with suicidal ideation during previous estrogen or ocp use.
* Known or suspected hypersensitivity to trial drug.
* Patients enrolled simultaneously into other investigative studies that require meds.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2007-08; Primary Completion 2011-03 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard S Legro, M.D., Principal Investigator — Penn State University
Locations (1):
- Nova Gradiska General Hospital, Strossmayerova 17, Croatia

REFERENCES:
- [Derived] Schroll JB, Black AY, Farquhar C, Chen I. Combined oral contraceptive pill for primary dysmenorrhoea. Cochrane Database Syst Rev. 2023 Jul 31;7(7):CD002120. doi: 10.1002/14651858.CD002120.pub4. PMID 37523477
- [Derived] Dmitrovic R, Kunselman AR, Legro RS. Continuous compared with cyclic oral contraceptives for the treatment of primary dysmenorrhea: a randomized controlled trial. Obstet Gynecol. 2012 Jun;119(6):1143-50. doi: 10.1097/AOG.0b013e318257217a. PMID 22617578

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Study Group (CCOCP) | Control Group (Traditional OCP)
Started | 19 | 19
Completed | 15 | 14
Not Completed | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Study Group (CCOCP) | Control Group (Traditional OCP) | Total
Number analyzed (Participants) | 19 | 19 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.47 (3.91) | 21.00 (4.03) | 20.74 (3.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 19 | 38
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Croatia | 19 | 19 | 38
BMI [Mean (Standard Deviation); unit: kg/m^2] | 21.20 (3.23) | 20.36 (1.77) | 20.78 (2.60)

OUTCOME MEASURES:

1. Primary Outcome: Change in Visual Analog Scale (VAS) Score
Description: Change in subjective perception of pain, as measured by the VAS. Subjects completed the VAS at baseline and 6 months. The VAS ranges from 0 (no pain) to 100 (worst pain). Therefore, a negative change in VAS indicates improvement in pain and a positive change in VAS indicates worsening of pain.
Time Frame: Baseline and 6 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Study Group (CCOCP) | Control Group (Traditional OCP)
Number analyzed (Participants) | 19 | 19
units on a scale | -74.8 [-86.1 to -63.5] | -58.7 [-70.3 to -47.2]
Statistical Analysis 1: Comparison: Study Group (CCOCP) vs Control Group (Traditional OCP); Test type: Superiority; p = 0.05, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Study Group (CCOCP) | Control Group (Traditional OCP)
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 0/19 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No